CLINICAL TRIAL: NCT04072848
Title: A Prospective Observational Cohort Study to Investigate the Physiological Agreement Between Arterial Sampling (the Reference Method) and Mathematically Arterialised Venous Blood
Brief Title: Mathematically Arterialised Testing of Hypercapnic Subjects Study
Acronym: MATHS
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: P02375
Record Dates: First submitted 2019-01-23; First posted 2019-08-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-05

CONDITIONS: Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational cohort study of patients admitted to hospital with suspected hypercapnic respiratory failure and requiring treatment with non-invasive ventilation (NIV) as part of standard, routine management. Contemporaneous blood gas samples will be obtained via arterial, capillary, and venous methods. The venous samples will undergo mathematical arterialisation via the v-TAC system. In line with standard medical care, arterial samples will be obtained before starting NIV and at two set points afterwards (day 1 post-NIV, and pre-discharge). Pre-existing clinical thresholds will be used to assess the reliability of v-TAC against ABG, the existing gold standard and will conduct a retrospective model of decision-making once the blood sampling component of the study is concluded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above.
* Admitted for consideration of home Non Invasive Ventilation.
* Due to undergo arterial blood gas sampling as part of routine clinical care

Exclusion Criteria:

* Inability to provide informed consent.
* Clinical necessity to perform blood gas sampling prior to allowing sufficient time for informed consent.
* Inability to obtain reliable SpO2 readings

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected chronic hypercapnic respiratory failure admitted as part of routine clinical care for consideration of home NIV.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in blood carbon dioxide level (PaCO2) | Between day 0 and day 1
  Change in PaCO2 between the pre-NIV (non-invasive ventilation) and day 1 NIV samples for ABG (arterial blood gas) versus v-TAC (arterialised venous blood gas)

SECONDARY OUTCOMES:
Change in PaCO2 between ABG versus v-TAC versus Capillary Blood Gas (CBG) versus Venous Blood Gas (VBG) | Between day 0 and day 1
  Change in PaCO2 between ABG versus v-TAC versus Capillary Blood Gas (CBG) versus Venous Blood Gas (VBG) between the pre-NIV and day 1 samples
Change in PaCO2 between ABG versus v-TAC versus Capillary Blood Gas (CBG) versus Venous Blood Gas (VBG) | Between day 0 and through to study completion, up to 3 days
  Change in PaCO2 between ABG versus v-TAC versus Capillary Blood Gas (CBG) versus Venous Blood Gas (VBG) between the pre-NIV and pre-discharge samples
Relative difficult in sampling | Between day 0 and through to study completion, up to 3 days
  Frequency of sampling error rate for ABG versus CBG versus VBG versus V-TAC
Patient experience | Between day 0 and through to study completion, up to 3 days
  Using Numeric Pain Scale where 0 is no pain, 5 is moderate pain and 10 is worst pain possible
Patient preference | Between day 0 and through to study completion, up to 3 days
  Patient preference for method of blood gas sampling will be recorded in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davies, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davies MG, Wozniak DR, Quinnell TG, Palas E, George S, Huang Y, Jayasekara R, Stoneman V, Smith IE, Thomsen LP, Rees SE. Comparison of mathematically arterialised venous blood gas sampling with arterial, capillary, and venous sampling in adult patients with hypercapnic respiratory failure: a single-centre longitudinal cohort study. BMJ Open Respir Res. 2023 Jun;10(1):e001537. doi: 10.1136/bmjresp-2022-001537. PMID 37369550